CLINICAL TRIAL: NCT04428281
Title: An Open-label, Multicenter Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of RO7248824 in Participants With Angelman Syndrome
Brief Title: A Study to Investigate the Safety, Tolerability, Pharmacokinetics (PK) and Pharmacodynamics (PD) of RO7248824 in Participants With Angelman Syndrome (AS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP41674; 2019-003787-48 (EudraCT Number); RG6091 (Other: RG Number)
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Angelman Syndrome
Keywords: RO7248824; Angelman; ASO; LNA; Angelman syndrome
MeSH Terms: conditions — Angelman Syndrome

STUDY DESIGN:
Intervention Model Description: Non-randomized, adaptive, open label, multiple ascending, intra-participant, dose-escalation study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (19):
- Cohort A1 RO7248824 (Experimental): Participants 5-12 years
  Interventions: Drug: RO7248824
- Cohort A2 RO7248824 (Experimental): Participants 5-12 years
  Interventions: Drug: RO7248824
- Cohort A3 RO7248824 (Experimental): Participants 5-12 years
  Interventions: Drug: RO7248824
- Cohort A4 RO7248824 (Experimental): Participants 5-12 years
  Interventions: Drug: RO7248824
- Cohort A5 RO7248824 (Experimental): Participants 5-12 years
  Interventions: Drug: RO7248824
- Cohort B1 RO7248824 (Experimental): Participants 1-4 years
  Interventions: Drug: RO7248824
- Cohort B2 RO7248824 (Experimental): Participants 1-4 years
  Interventions: Drug: RO7248824
- Cohort B3 RO7248824 (Experimental): Participants 1-4 years
  Interventions: Drug: RO7248824
- Cohort B4 RO7248824 (Experimental): Participants 1-4 years
  Interventions: Drug: RO7248824
- Cohort B5 RO7248824 (Experimental): Participants 1-4 years
  Interventions: Drug: RO7248824
- LTE: Cohort EA1 RO7248824 (Experimental): New participants (age 5-12) enrolling directly in the LTE part
  Interventions: Drug: RO7248824
- LTE: Cohort EA2 RO7248824 (Experimental): Participants continuing from multiple ascending dose (MAD) cohorts A1 and A2
  Interventions: Drug: RO7248824
- LTE: Cohort EA3 RO7248824 (Experimental): Participants continuing from MAD cohorts A3 and A4
  Interventions: Drug: RO7248824
- LTE: Cohort EA4 RO7248824 (Experimental): Participants continuing from MAD Cohort A5
  Interventions: Drug: RO7248824
- LTE: Cohort EB1 RO7248824 (Experimental): New participants (age 1-4) enrolling directly into the LTE
  Interventions: Drug: RO7248824
- LTE: Cohort EB2 RO7248824 (Experimental): Participants continuing from MAD cohorts B1 and B2
  Interventions: Drug: RO7248824
- LTE: Cohort EB3 RO7248824 (Experimental): Participants continuing from MAD cohorts B3 and B4
  Interventions: Drug: RO7248824
- LTE: Cohort EB4 RO7248824 (Experimental): Participants continuing from MAD Cohort B5
  Interventions: Drug: RO7248824
- OOE: RO7248824 (Experimental): Participants in the LTE part of the study will be given the opportunity to participate in the OOE part.
  Interventions: Drug: RO7248824

INTERVENTIONS:
Drug: RO7248824 — In the MAD part, RO7248824 will be administered as IT injection of varing dose levels over a period of 8 weeks, with a minimum of approximately 4 weeks between each dose administration. In the LTE part, RO7248824 will be administered as IT injection of varying dose levels over a period of 144 weeks, with a minimum of approximately 16 weeks between each dose administration. In the OOE part, participants will receive RO7248824 as an IT injection with the same dosing regime as the LTE part over a period of up to 48 weeks.

SUMMARY:
This is a phase I, multicenter, non-randomized, adaptive, open-label, multiple ascending, intra-participant, dose-escalation study with a long-term extension (LTE) part and an optional open-label extension (OOE) part. The objective of the study is to investigate the safety, tolerability, PK and PD of RO7248824 administered intrathecally (IT) in participants with AS. Two linked sets of dose escalation cohorts are planned based on two different age groups, namely participants with AS aged ≥ 5 to ≤ 12 years in cohorts A1 to A5 (with at least 2 participants ≤ 8 years old in each cohort) and AS participants aged ≥ 1 to ≤ 4 years in cohorts B1 to B5. The two sets of cohorts will be run in parallel, with each cohort A1 to A5 preceding and gating the linked cohort B1 to B5 (e.g., A1 precedes B1).

ELIGIBILITY:
Inclusion Criteria:

* The participant has a parent, caregiver or legal representative (hereinafter "caregiver") who is reliable, competent and at least 18 years of age. The caregiver is willing and able to accompany the participant to clinic visits and to be available to the Investigational Site by phone or email if needed and who (in the opinion of the Investigator) is and will remain sufficiently knowledgeable of participant's ongoing condition to respond to any inquiries about the participant from personnel from the Study Site.
* A caregiver must be able to consent for the participant according to International Council on Harmonisation (ICH) and local regulations.
* Ability to comply with all study requirements.
* Have adequate supportive psychosocial circumstances.
* Able to tolerate blood draws.
* Able to undergo lumbar puncture (LP) and IT injection, under sedation or anesthesia if needed and as determined appropriate by the Investigator.
* Stable medical status for at least 4 weeks prior to Screening and at the time of enrollment.
* Body weight of ≥ 7 kg
* Participant must be ≥ 1 to ≤ 12 years of age at the time of signing of the informed consent by the caregiver.
* Clinical diagnosis of AS confirmed by a molecular diagnosis with genotypic classification of either Ubiquitin-protein ligase E3A (UBE3A) mutation of the maternal allele or deletion on the maternally inherited chromosome 15q11q13 that includes the UBE3A gene and is less than 7 megabyte (Mb) in size.

Reproductive Status:

Some of the provisions that follow may have limited applicability based on the age range of study participants (i.e., up to the age of 12) and the nature of the disease understudy. These provisions are nonetheless included for purposes of completeness in order:

A) Female Participants

A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

* Women of non-childbearing potential.
* Women of childbearing potential who agree to remain abstinent (refrain from heterosexual intercourse) or use acceptable contraceptive methods during the treatment period and for at least 6 months after the final dose of RO7248824 (RG6091). The following are acceptable contraceptive methods: bilateral tubal occlusion/ ligation, male sexual partner who is sterilized, established proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices and copper intrauterine devices, male or female condom with or without spermicide; and cap, diaphragm, or sponge with spermicide.

B) Male Participants

During the treatment period and for at least 6 months after the final dose of RO7248824 (RG6091), consent has to be provided to:

* Remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures such as a condom, with a female partner of childbearing potential, or pregnant female partner, to avoid exposing the embryo.

The reliability of sexual abstinence for male and/or female enrollment eligibility needs to be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the participant. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not acceptable methods of preventing drug exposure.

Inclusion Criteria for OOE Part:

- Current or prior participations in the LTE part of Study BP41674.

Exclusion Criteria:

Diagnostic Assessments

* Clinically-significant laboratory, vital sign or electrocardiography (ECG) abnormalities at Screening

Type of Participants and Disease Characteristics

* Molecular diagnosis of AS with genotypic classification: Paternal Uniparental Disomy (UPD) of 15q11-13; UBE3A Imprinting center defect (ID); A partial molecular diagnosis of AS, that cannot exclude (UPD)or ID despite appropriate genetic testing.
* Clinically relevant hematological, hepatic, cardiac or renal disease or event, in the judgement of the Investigator.
* Any concomitant condition that might interfere with the clinical evaluation of AS and that is not related to AS.
* Known history of human immunodeficiency virus (HIV) or hepatitis B virus (HBV) or hepatitis C virus (HCV).
* Any condition that increases risk of meningitis.
* History of bleeding diathesis or coagulopathy.
* A medical history of brain or spinal disease that would interfere with the LP process, CSF circulation or safety assessment
* History of clinically significant post-lumbar-puncture headache of moderate or severe intensity and/or blood patch
* Malignancy within 5 years of Screening
* Hospitalization for any major medical or surgical procedure involving general anesthesia within 12 weeks of Screening or planned during the study
* Have any other conditions, which, in the opinion of the Investigator, would make the participant unsuitable for inclusion or could interfere with the participant participating in or completing the study, including any contraindication to administration of intrathecal therapy.
* Premature birth with gestational age at birth below 34 weeks.
* History of hypersensitivity to the investigational medicinal product (IMP), antisense oligonucleotides, or any excipients.

Prior Therapy

* Allowed sleep medications have not been stable for 4 weeks prior to screening and at the time of enrollement.
* Allowed medications for treatment of epilepsy have not been stable for 12 weeks prior to screening and at the time of enrollment.
* Use of antiplatelet or anticoagulant therapy for 2 weeks prior to screening and at the time of enrollment.
* Concurrent psychotropic medications have not been stable for 4 weeks prior to screening and at the time of enrollment.

Other Exclusion Criteria: Prior/Concurrent Clinical Study Experience

* Received an investigational drug within 90 days or 5 times the half-life of the investigational drug (whichever is longer) or participation in a study testing an investigational medical device within 90 days prior to first dosing or if the device is still active.
* Concurrent or planned concurrent participation in any clinical study (including observational, non-drug and non-interventional studies) without a signed data sharing agreement in place between the other clinical study and the Sponsor.
* Previous participation in a cellular therapy, or gene therapy, or gene editing clinical study.

Exclusion Criteria for OOE Part:

- Participants who never enrolled in Study BP41674, or who discontinued participation due to safety reasons, are not eligible for the OOE part.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Frequency and Severity of Adverse Events (AEs) | Baseline to last visit or early withdrawal
  MAD part: From the baseline MAD visit to the final MAD visit (Day 365) or early withdrawal.
  LTE part: From the baseline LTE visit to final LTE visit (Day 1092) or early withdrawal.
  OOE part: From baseline OOE visit to final OOE visit (Day 420) or early termination.
Frequency and Severity of Serious Adverse Events (SAEs) | Baseline to last visit or early withdrawal
  MAD part: From the baseline MAD visit to the final MAD visit (Day 365) or early withdrawal.
  LTE part: From the baseline LTE visit to final LTE visit (Day 1092) or early withdrawal.
  OOE part: From baseline OOE visit to final OOE visit (Day 420) or early termination.
Number of Participants Discontinued Treatment due to AEs | Baseline to last visit or early withdrawal
  MAD part: From the baseline MAD visit to the final MAD visit (Day 365) or early withdrawal.
  LTE part: From the baseline LTE visit to final LTE visit (Day 1092) or early withdrawal.
  OOE part: From baseline OOE visit to final OOE visit (Day 420) or early termination.
Frequency of Abnormal Laboratory Findings (Blood, Cerebrospinal Fluid [CSF] and Urinalysis) | Baseline to last visit or early withdrawal
  MAD part: From the baseline MAD visit to the final MAD visit (Day 365) or early withdrawal.
  LTE part: From the baseline LTE visit to final LTE visit (Day 1092) or early withdrawal.
  OOE part: From baseline OOE visit to final OOE visit (Day 420) or early termination.
Frequency of Abnormal Vital Signs | Baseline to last visit or early withdrawal
  MAD part: From the baseline MAD visit to the final MAD visit (Day 365) or early withdrawal.
  LTE part: From the baseline LTE visit to final LTE visit (Day 1092) or early withdrawal.
Frequency of Abnormal Electrocardiography (ECG) Values | Baseline to last visit or early withdrawal
  MAD part: From the baseline MAD visit to the final MAD visit (Day 365) or early withdrawal.
  LTE part: From the baseline LTE visit to final LTE visit (Day 1092) or early withdrawal.
Mean Changes From Baseline in Temperature Over Time | Baseline to last visit or early withdrawal
  MAD part: From the baseline MAD visit to the final MAD visit (Day 365) or early withdrawal.
  LTE part: From the baseline LTE visit to final LTE visit (Day 1092) or early withdrawal.
Mean Changes From Baseline in Systolic Blood Pressure Over Time | Baseline to last visit or early withdrawal
  MAD part: From the baseline MAD visit to the final MAD visit (Day 365) or early withdrawal.
  LTE part: From the baseline LTE visit to final LTE visit (Day 1092) or early withdrawal.
Mean Changes From Baseline in Diastolic Blood Pressure Over Time | Baseline to last visit or early withdrawal
  MAD part: From the baseline MAD visit to the final MAD visit (Day 365) or early withdrawal.
  LTE part: From the baseline LTE visit to final LTE visit (Day 1092) or early withdrawal.
Mean Changes From Baseline in Heartrate Over Time | Baseline to last visit or early withdrawal
  MAD part: From the baseline MAD visit to the final MAD visit (D365) or early withdrawal.
  LTE part: From the baseline LTE visit to final LTE visit (D1092) or early withdrawal.
Mean Changes From Baseline in Respiratory Rate Over Time | Baseline to last visit or early withdrawal
  MAD part: From the baseline MAD visit to the final MAD visit (Day 365) or early withdrawal.
  LTE part: From the baseline LTE visit to final LTE visit (Day 1092) or early withdrawal.

SECONDARY OUTCOMES:
Time to Maximum Concentration (Tmax) for RO7248824 | Baseline to last visit or early withdrawal
  MAD part: From the baseline MAD visit to the final MAD visit (Day 365) or early withdrawal.
  LTE part: From the baseline LTE visit to final LTE visit (Day 1092) or early withdrawal.
Maximum Plasma Concentration Observed (Cmax) for RO7248824 | Baseline to last visit or early withdrawal
  MAD part: From the baseline MAD visit to the final MAD visit (Day 365) or early withdrawal.
  LTE part: From the baseline LTE visit to final LTE visit (Day 1092) or early withdrawal.
Area Under Curve (AUC) From Time 0 to Time of Last Sampling Point or Last Quantifiable Sample, Whichever Comes First (AUC last) for RO7248824 | Baseline to last visit or early withdrawal
  MAD part: From the baseline MAD visit to the final MAD visit (Day 365) or early withdrawal.
  LTE part: From the baseline LTE visit to final LTE visit (Day 1092) or early withdrawal.
AUC From Time 0 to Infinity (AUCinf) for RO7248824 | Baseline to last visit or early withdrawal
  MAD part: From the baseline MAD visit to the final MAD visit (Day 365) or early withdrawal.
  LTE part: From the baseline LTE visit to final LTE visit (Day 1092) or early withdrawal.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (12):
- United States (7):
  - UCLA Neuropsychiatric Institute, Los Angeles, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Rush Medical Center, Chicago, Illinois
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Columbia University Medical Center, New York, New York
  - Carolina Institute for Development DisabilitiesUniversity of North Carolina/School of Medicine, Carrboro, North Carolina
  - Baylor College of Med, Houston, Texas
- Ospedale Pediatrico Bambino Gesù, Rome, Lazio, Italy
- Erasmus MC / location Sophia Kinderziekenhuis, Rotterdam, Netherlands
- Spain (3):
  - Hospital Sant Joan De Deu, Esplugues de Llobregas, Barcelona
  - Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona
  - Hospital Universitario Virgen del Rocío, Seville

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/members/ourmembers/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Hipp JF, Bacino CA, Bird LM, Bruenig-Traebert I, Chan D, de Wit MC, Fontoura P, Hooper G, Jagasia R, Krishnan ML, Murtagh L, Noci A, Martinez AR, Schwab D, Serrano M, Shen MD, Tillmann J, Tjeertes J, Vincenzi B, Berry-Kravis E, Bonni A; Rugonersen Study Group; all TANGELO investigators. The UBE3A-ATS antisense oligonucleotide rugonersen in children with Angelman syndrome: a phase 1 trial. Nat Med. 2025 Sep;31(9):2936-2945. doi: 10.1038/s41591-025-03784-7. Epub 2025 Jul 11. PMID 40646322